CLINICAL TRIAL: NCT01351441
Title: Minimizing Risk and Maximizing Outcomes in Geriatric Patients Through Integrated Clinical Pharmacy Services in an Innovative Model of Community Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VascuScript Pharmacy (Other)
Collaborators: Community Pharmacy Foundation (Other)
Responsible Party: Principal Investigator, Scott V. Monte, Clinical Assistant Professor, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PHP1140411E
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Medication Adherence; Health Literacy; Geriatric Patient Care Improvement; Pharmacy Economic Improvement
Keywords: Geriatric; Pharmacoeconomics; Health Literacy; Adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Age 65 years or over AND at least 5 chronic medications (Other)
  Interventions: Behavioral: Medication adherence consultation; Other: Medication problems assessment; Other: Beer's Criteria Assessment; Behavioral: Health Literacy Assessment

INTERVENTIONS:
Behavioral: Medication adherence consultation — Patients will be counseled in person on day 0 then telephonically every month after until day 365.
Other: Medication problems assessment — Patients will be asked if they are having any issues that may be attributable to their current drug therapy on a monthly basis. Any issue that is identified will be addressed by the pharmacist.
Other: Beer's Criteria Assessment — The patient's drug therapy will be reviewed for Beer's criteria medications and possible alternatives will be addressed by the pharmacist if deemed appropriate.
Behavioral: Health Literacy Assessment — Patients will be given a Health Literacy Assessment on day 0 and day 365 using the Realm-SF.

SUMMARY:
It has been shown that patients can improve their safety through informed choice, safe medication use, and complication reporting. This includes not only the potential problems that occur from prescription medication use but also issues that may arise through the improper use of over-the-counter medications. The willingness of a patient to take on safety action is known to be complicated by an unwillingness to behave in a manner that might challenge a physician's judgment or actions. Community pharmacists are in the unique position to provide perspective on the physician's recommendation and act as an advocate to facilitate necessary change. Through supportive and repeated interaction with their community pharmacist patients will develop assertiveness toward their own health care, an increased frequency and quality of interaction with their physician, and thus a minimized risk of harm and maximized opportunity to optimize clinical outcomes.

DETAILED DESCRIPTION:
This is a single center, observational study to determine if geriatric patients who are on five or more chronic medications will have a difference in clinical, humanistic, and/or economic outcome through an integrated clinical pharmacy service intervention. The primary efficacy objective will be assessed through a single cohort, paired research design measuring the change from baseline in the adherence rate, number of medication related problems, and Beers criteria medications. The primary economic objective will be assessed through prescription revenue to validate the employment of a 0.5-1.0 Full-time equivalent (FTE). Secondary efficacy objectives will be assessed through a single cohort, paired research design measuring the change from baseline in the health literacy, optimization in the anthropometrics, and health related quality of life (HRQOL).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least 65 years of age
* Have at least 5 medications that they take on a chronic basis
* Willing to have their prescriptions filled by VascuScript Pharmacy
* Understand the terms of the informed consent

Exclusion Criteria:

* Any patient who does not meet the requirements of the Inclusion Criteria

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Medication adherence | Every 30 days for 12 months
  To determine if an integrated clinical pharmacy service program in geriatric patients can maintain a medication adherence rate ≥80%.
Medication related problems | Every 30 days for 12 months
  To determine if an integrated clinical pharmacy service program in geriatric patients can reduce the number of medication related problems by ≥10%.
Beers criteria medications | Every month for 12 months
  To determine if an integrated clinical pharmacy service program in geriatric patients can reduce the number of Beers criteria medications by ≥10%.
Economic impact | 12 months
  To determine the number of patients required to validate a part-time or full-time pharmacist to perform the required clinical functions of the clinical pharmacy service geriatric program.

SECONDARY OUTCOMES:
Health literacy | 12 months
  To determine if an integrated clinical pharmacy service program in geriatric patients can improve health literacy as evidenced by the REALM-SF.
Optimizing Anthropometrics | 12 months
  To determine if an integrated clinical pharmacy service program in geriatric patients can demonstrate ≥10% improvement and/or greater optimization of patient weight, blood pressure, cholesterol, and blood glucose (if applicable).
Quality of Life | 12 months
  To determine if an integrated clinical pharmacy service program in geriatric patients can improve quality of life as evidenced by the CDC HRQOL Healthy Days Core Module.

CONTACTS AND LOCATIONS:
Locations (1):
- VascuScript Pharmacy, Cheektowaga, New York, United States